CLINICAL TRIAL: NCT03042078
Title: Multi-center, Controlled Trial to Compare the Feasibility, Safety and Efficacy of Zero-fluoroscopic Approach With Fluoroscopic Approach for the Ablation of Paroxysmal Supraventricular Tachycardia
Brief Title: Zero-fluoroscopy Approach Versus Fluoroscopic Approach for the Ablation of Paroxysmal Supraventricular Tachycardia
Acronym: ZFA-PSVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Xiangyang Central Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Guangdong Provincial People's Hospital (Other); Morristown Memorial Hospital (Other); Beijing Anzhen Hospital (Other); Ningbo No. 1 Hospital (Other)
Responsible Party: Principal Investigator, Yan Wang, Professor, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJHCDD-ZF-PSVT-20140301
Record Dates: First submitted 2017-01-27; First posted 2017-02-03 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Paroxysmal Supraventricular Tachycardia
Keywords: Fluoroscopy; Ablation; Three dimensional; Paroxysmal supraventricular tachycardia; Radiation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zero-fluoroscopic ablation (Experimental): Paroxysmal supraventricular tachycardia will be ablated under the guidance of Ensite NavX and without the use of fluoroscopy.
  Interventions: Device: Zero-fluoroscopic ablation
- Conventional fluoroscopic ablation (Active Comparator): Paroxysmal supraventricular tachycardia will be ablated under the guidance of Ensite NavX plus fluoroscopy.
  Interventions: Device: Conventional fluoroscopic ablation

INTERVENTIONS:
Device: Zero-fluoroscopic ablation — Catheter ablation will be performed under the guidance of Ensite NavX and without the use of fluoroscopy.
  Arms: Zero-fluoroscopic ablation
Device: Conventional fluoroscopic ablation — Catheter ablation will be performed under the guidance of Ensite NavX plus fluoroscopy.
  Arms: Conventional fluoroscopic ablation

SUMMARY:
This study is aimed to compare the feasibility, safety and efficacy of a zero-fluoroscopic approach using Ensite NavX with conventional fluoroscopic approach using Ensite NavX plus fluoroscopy for the ablation of paroxysmal supraventricular tachycardia.

DETAILED DESCRIPTION:
Fluoroscopy is the imagine modality routinely used in catheter ablation of cardiac arrhythmias. As we all know,fluoroscopic radiation is harmful both to the patients and the operation staffs. Recently,three-dimensional navigation systems have been developed and implemented in electrophysiological procedures for guiding catheters inside the heart chambers. Among the three-dimensional navigation systems, Ensite NavX is a promising system used for zero-fluoroscopic approach for performing catheter ablation of paroxysmal supraventricular tachycardia. This study is aimed to compare the feasibility, safety and efficacy of a zero-fluoroscopic approach using Ensite NavX with conventional fluoroscopic approach using Ensite NavX plus fluoroscopy for the ablation of paroxysmal supraventricular tachycardia.

ELIGIBILITY:
Inclusion Criteria:

* Atrioventricular Nodal Reentrant Tachycardia
* Atrioventricular Reentrant Tachycardia

Exclusion Criteria:

* Atrial Tachycardia
* Organic supraventricular tachycardia

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3060 (Actual)
Dates: Start 2012-01; Primary Completion 2018-02 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Procedural success rate | one year
  Procedural success for AVNRT was defined as the absence of inducible tachycardia either under basal condition or under isoproterenol stimulation. Procedural success for AVRT was defined as the non-inducibility of tachycardia, loss of pre-excitation (if manifest), loss of retrograde accessory pathway conduction and transient atrioventricular block induced by intravenous adenosine.

SECONDARY OUTCOMES:
Complications | one year
  Complications were defined as pseudoaneurysm, arterialvenous fistula, pneumothorax, second- or third-degree atrioventricular block, cardiac tamponade, or other serious complications requiring intervention.
Immediate success rate | one day
  Procedural success for AVNRT was defined as the absence of inducible tachycardia either under basal condition or under isoproterenol stimulation. Procedural success for AVRT was defined as the non-inducibility of tachycardia, loss of pre-excitation (if manifest), loss of retrograde accessory pathway conduction and transient atrioventricular block induced by intravenous adenosine.
Recurrence Rate | 1 year
  2. An ECG and electrophysiology study would be performed to rule out recurrence when the patients had suspicious symptoms or signs.
Total procedure time | one day
  Procedure time (in minutes) was defined as the interval from the beginning of local anesthesia to extraction of all femoral venous sheaths at the end of the procedure. Total ablation time was calculated in seconds but time for tentative ablation was not taken into account.
Fluoroscopy time | one day
  2. Fluoroscopy time (in minutes) was defined as thetotal duration of exposure during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, PhD, Principal Investigator — Tongji Hospital Wuhan, Hubei China
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anselmino M, Sillano D, Casolati D, Ferraris F, Scaglione M, Gaita F. A new electrophysiology era: zero fluoroscopy. J Cardiovasc Med (Hagerstown). 2013 Mar;14(3):221-7. doi: 10.2459/JCM.0b013e3283536555. PMID 22526222
- [Background] Mobinizadeh M, Arabloo J, Hamouzadeh P, Akbari Sari A. A systematic review of the effectiveness of catheter ablation NavX mapping system for treatment of the cardiac arrhythmia. Med J Islam Repub Iran. 2015 Mar 10;29:189. eCollection 2015. PMID 26034742
- [Background] Wang Y, Patel D, Wang DW, Yan JT, Hsia HH, Liu H, Zhao CX, Zuo HJ, Wang DW. beta1-Adrenoceptor blocker aggravated ventricular arrhythmia. Pacing Clin Electrophysiol. 2013 Nov;36(11):1348-56. doi: 10.1111/pace.12196. Epub 2013 Jun 10. PMID 23750689
- [Background] Lim PB, Robb D, Lambiase PD. Electrophysiology and ablation of arrhythmias. Br J Hosp Med (Lond). 2012 Jun;73(6):312-8. doi: 10.12968/hmed.2012.73.6.312. PMID 22875320
- [Background] Brown KR, Rzucidlo E. Acute and chronic radiation injury. J Vasc Surg. 2011 Jan;53(1 Suppl):15S-21S. doi: 10.1016/j.jvs.2010.06.175. Epub 2010 Sep 16. PMID 20843630
- [Derived] Chen G, Wang Y, Proietti R, Wang X, Ouyang F, Ma CS, Yu RH, Zhao C, Ma K, Qiu J, Liu Q, Wang DW. Zero-fluoroscopy approach for ablation of supraventricular tachycardia using the Ensite NavX system: a multicenter experience. BMC Cardiovasc Disord. 2020 Feb 3;20(1):48. doi: 10.1186/s12872-020-01344-0. PMID 32013865